CLINICAL TRIAL: NCT02270736
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study With an Open-label Extension Period to Investigate the Efficacy and Safety of NT 201 in the Treatment of Children and Adolescents (2-17 Years) With Chronic Troublesome Sialorrhea Associated With Neurological Disorders, and/or Intellectual Disability
Brief Title: Clinical Study to Investigate the Efficacy and Safety of NT 201 Compared to Placebo in the Treatment of Chronic Troublesome Drooling Associated With Neurological Disorders and/or Intellectual Disability
Acronym: SIPEXI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ60201_3091_1; 2013-004532-30 (EudraCT Number)
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Troublesome Sialorrhea; Cerebral Palsy; Stroke; Traumatic Brain Injury; Intellectual Disability
MeSH Terms: conditions — Cerebral Palsy; Stroke; Brain Injuries, Traumatic; Intellectual Disability | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind MP: Placebo (Age 6 to 17 Years) (Experimental): Participants will receive placebo via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks. Volumes will be matched to the volumes of NT 201 (incobotulinumtoxinA; Xeomin) injected in the experimental arm.
  Interventions: Drug: NT 201 Placebo
- Double-blind, MP: NT 201 (Age 6 to 17 Years) (Experimental): Participants will receive NT 201 (up to 2.5 Units per kilogram [U/kg] body weight) via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks.
  Interventions: Drug: NT 201
- Open-label, MP: NT 201 (Age 2 to 5 Years) (Experimental): Participants will receive NT 201 (about 1.5-2 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks.
  Interventions: Drug: NT 201
- OLEX: NT 201 (Age 6 to 17 Years) (Experimental): Participants will receive NT 201 (up to 2.5 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 of second (Visit 6), third (Visit 10), and fourth (Visit 14) injection cycle of the OLEX, followed by an observation period of 16 weeks each (48 weeks in total). This arm will consist of participants who will participate in MP arms "Double-blind, MP: placebo (age 6 to 17 years)" and "Double-blind, MP: NT 201 (age 6 to 17 years)".
  Interventions: Drug: NT 201
- OLEX: NT 201 (Age 2 to 5 Years) (Experimental): Participants will receive NT 201 (about 1.5-2 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 of second (Visit 6), third (Visit 10), and fourth (Visit 14) injection cycle of the OLEX, followed by an observation period of 16 weeks each (48 weeks in total).
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 Placebo — NT 201 placebo matching injection.
  Arms: Double-blind MP: Placebo (Age 6 to 17 Years)
Drug: NT 201 — NT 201 injection.
  Other Names: IncobotulinumtoxinA; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: Double-blind, MP: NT 201 (Age 6 to 17 Years); OLEX: NT 201 (Age 2 to 5 Years); OLEX: NT 201 (Age 6 to 17 Years); Open-label, MP: NT 201 (Age 2 to 5 Years)

SUMMARY:
The objective of this study is to investigate the efficacy and safety of NT 201 compared with placebo for the treatment of chronic troublesome sialorrhea associated with neurological disorders (e.g. cerebral palsy, traumatic brain injury) and/or intellectual disability in children and adolescents naïve to Botulinum neurotoxin treatment and aged 2-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child/adolescent age 2-17 years.
* Any neurological disorder (e.g. cerebral palsy or traumatic brain injury) and/or intellectual disability associated with chronic troublesome sialorrhea for at least 3 months up to the screening. In subjects with intellectual disability (ID) without neurological disorders, a diagnosis of ID by a specialist, e.g. pediatrician or by a center for developmental medicine is required for inclusion.
* Severe drooling (modified Teacher´s Drooling Scale [mTDS] ≥ 6; clothing occasionally becomes damp) as rated by the investigator.
* Parental consent and the subject's oral or written assent as the subject is able to provide.

Exclusion Criteria:

* Chronic troublesome sialorrhea not related to neurological disorders and/or intellectual disability.
* Body weight < 12 kg.
* Pharmacological treatment for sialorrhea or concomitant medication known to influence sialorrhea strongly (e.g. anticholinergics with exception of locally applied or short acting drugs used under general anesthesia) within 45 days before baseline and during the entire study period.
* Any previous known or suspected hypersensitivity to Botulinum toxin.
* Aspiration pneumonia within 6 month before screening.
* Any previous treatment with Botulinum toxin for any body region during the year before screening or within the screening period
* Prior, concomitant or planned surgery or irradiation to head and neck to control sialorrhea (including salivary gland surgery or salivary gland irradiation) within one year before screening or planned for any part of the entire study period.
* Concurrent diseases, including hematological, hepatic, renal, gastrointestinal, endocrine, pulmonary, musculoskeletal, or psychiatric diseases or conditions, which in the judgment of the investigator would put the subject at risk while in the study, could influence the results of the study, or negatively impact the subject's ability to participate in the study.
* Extremely poor dental and/or oral condition that might preclude safe study participation by the judgment of the investigator.
* Nursing mother or pregnant female subject.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (31):
- Georgia (3):
  - Merz Investigational Site #9950003, K'obulet'i
  - Merz Investigational Site #9950001, Tbilisi
  - Merz Investigational Site #9950002, Tbilisi
- Hungary (6):
  - Merz Investigational Site #0360017, Balassagyarmat
  - Merz Investigational Site #0360013, Budapest
  - Merz Investigational Site # 0360014, Budapest
  - Merz Investigational Site # 0360015, Budapest
  - Merz Investigational Site #0360018, Budapest
  - Merz Investigational Site #0360016, Szombathely
- Poland (5):
  - Merz Investigational Site #0480092, Bialystok
  - Merz Investigational Site #0480090, Gdansk
  - Merz Investigational Site #0480076, Katowice
  - Merz Investigational Site #0480059, Krakow
  - Merz Investigational Site #0480060, Wiązowna
- Russia (8):
  - Merz Investigational Site #0070016, Kazan'
  - Merz Investigational Site # 0070288, Kemerovo
  - Merz Investigational Site #0070290, Khabarovsk
  - Merz Investigational # 0070017, Saint Petersburg
  - Merz Investigational Site #0070013, Smolensk
  - Merz Investigational Site # 070019, Stavropol
  - Merz Investigational Site #0070300, Tomsk
  - Merz Investigational Site #0070301, Yekaterinburg
- Merz Investigational Site #3810001, Belgrade, Serbia
- Ukraine (8):
  - Merz Investigational Site #3800001, Dnipropetrovsk
  - Merz Investigational Site #3800012, Ivano-Frankivsk
  - Merz Investigational Site #3800005, Kharkiv
  - Merz Investigational Site #3800007, Kharkiv
  - Merz Investigational Site #3800013, Kherson
  - Merz Investigational site #3800003, Odesa
  - Merz Investigational Site #3800009, Ternopil
  - Merz Investigational Site #3800011, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berweck S, Bonikowski M, Kim H, Althaus M, Flatau-Baque B, Mueller D, Banach MD. Placebo-Controlled Clinical Trial of IncobotulinumtoxinA for Sialorrhea in Children: SIPEXI. Neurology. 2021 Oct 4;97(14):e1425-e1436. doi: 10.1212/WNL.0000000000012573. PMID 34341153
- [Derived] Berweck S, Banach M, Gaebler-Spira D, Chambers HG, Schroeder AS, Geister TL, Althaus M, Hanschmann A, Vacchelli M, Bonfert MV, Heinen F, Dabrowski E. Safety Profile and Lack of Immunogenicity of IncobotulinumtoxinA in Pediatric Spasticity and Sialorrhea: A Pooled Analysis. Toxins (Basel). 2022 Aug 25;14(9):585. doi: 10.3390/toxins14090585. PMID 36136523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 investigational sites in Georgia, Hungary, Poland, Russia, Serbia, and Ukraine.
Pre-assignment Details: A total of 281 participants were screened, out of which 256 participants were enrolled/randomized into the study. Of these 256 participants, 255 participants received the study treatment. A total of 247 participants who completed the Main Period (MP) entered the Open-label Extension Period (OLEX) of the study.
Groups:
- Double-blind MP: Placebo (Age 6 to 17 Years): Participants received placebo via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks. Volumes were matched to the volumes of NT 201 (incobotulinumtoxinA; Xeomin) injected in the experimental arm.
- Double-blind, MP: NT 201 (Age 6 to 17 Years): Participants received NT 201 (up to 2.5 Units per kilogram [U/kg] body weight) via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks.
- Open-label, MP: NT 201 (Age 2 to 5 Years): Participants received NT 201 (about 1.5-2 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks.
- OLEX: NT 201 (Age 6 to 17 Years): Participants received NT 201 (up to 2.5 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 of second (Visit 6), third (Visit 10), and fourth (Visit 14) injection cycle of the OLEX, followed by an observation period of 16 weeks each (48 weeks in total). This arm consisted of participants who participated in MP arms "Double-blind, MP: placebo (age 6 to 17 years)" and "Double-blind, MP: NT 201 (age 6 to 17 years)".
- OLEX: NT 201 (Age 2 to 5 Years): Participants received NT 201 (about 1.5-2 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 of second (Visit 6), third (Visit 10), and fourth (Visit 14) injection cycle of the OLEX, followed by an observation period of 16 weeks each (48 weeks in total).
Period: Main Period (MP) (up to 16 Weeks)
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Started | 72 | 148 | 36 | 0 | 0
Treated | 72 | 148 | 35 | 0 | 0
Completed | 70 | 146 | 34 | 0 | 0
Not Completed | 2 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Randomized, not Treated | 0 | 0 | 1 | 0 | 0
Period: OLEX Period (up to 48 Weeks)
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Started | 0 | 0 | 0 | 214 (2 participants from MP did not enter OLEX due to withdrawal of consent.) | 33 (1 participant from MP did not enter OLEX due to adverse event.)
Completed | 0 | 0 | 0 | 189 | 33
Not Completed | 0 | 0 | 0 | 25 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 16 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety evaluable set (SES) (MP) is the subset of all participants who received study medication (NT 201 or placebo) during the MP of the study.
Groups:
- Double-blind, MP: NT 201 (Age 6 to 17 Years): Participants received NT 201 (up to 2.5 U/kg body weight) via bilateral intraglandular injection into the parotid and submandibular glands in one injection session on Day 1 (Visit 2) of the MP, followed by an observation period of 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | Total
Number analyzed (Participants) | 72 | 148 | 35 | 255
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0
  Children (2-11 years) | 48 | 96 | 35 | 179
  Adolescents (12-17 years) | 24 | 52 | 0 | 76
  Adults (18-64 years) | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 55 | 13 | 95
  Male | 45 | 93 | 22 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 72 | 148 | 35 | 255
  Black or African American | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 135.3 (16.92) | 132.8 (17.15) | 101.1 (8.09) | 129.1 (19.64)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 30.8 (11.67) | 28.8 (11.48) | 15.7 (3.00) | 27.6 (11.78)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 16.4 (3.65) | 15.8 (3.25) | 15.3 (1.85) | 15.9 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unstimulated Salivary Flow Rate (uSFR) at Week 4
Description: This endpoint was planned to be analyzed in double-blind, MP, 6 to 17 years participants only. uSFR was assessed by weighing of absorbent swabs with safety threads soaked with saliva over 5 minutes and the procedure was repeated after 30 minutes. Salivary flow rate was equal to weight increase of swabs/time of collection. The average of the 2 results for flow rate was calculated. The reduction of measured weight over the study relates to improvement of sialorrhea.
Time Frame: Baseline and Week 4
Population: The full analysis set (FAS) is identical to the subset of participants in the SES (MP) where subset of all participants received study medication (NT 201 or placebo) during the MP of the study.
Measure: Least Squares Mean (Standard Error); unit: gram per minute (g/min)
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years)
Number analyzed (Participants) | 72 | 148
gram per minute (g/min) | -0.07 (0.015) | -0.14 (0.012)
Statistical Analysis 1: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); Least square mean (LS-Mean) is from a mixed model repeated measurement (MMRM) analysis with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline uSFR score as covariate; Test type: Superiority; p = 0.0012, MMRM; Least square mean (LS-mean) difference = -0.06, 95% CI 2-sided [-0.1 to -0.03], Standard Error of Mean 0.019

2. Primary Outcome: Global Impression of Change Scale (GICS) at Week 4 Assessed by the Carer/Parent(s)
Description: This endpoint was analyzed in double-blind, MP, 6 to 17 years participants. The GICS was used to measure the carer's/parent's impression of change due to treatment. The response option was a common 7-point Likert scale, with the following values: +3 (very much improved); +2 (much improved); +1 (minimally improved); 0 (no change); -1 (minimally worse); -2 (much worse); -3 (very much worse).
Time Frame: Week 4
Population: The FAS is identical to the subset of participants in the SES (MP) where subset of all participants received study medication (NT 201 or placebo) during the MP of the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years)
Number analyzed (Participants) | 72 | 148
units on a scale | 0.63 (0.104) | 0.91 (0.075)
Statistical Analysis 1: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); LS-Mean is from a MMRM analysis model with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline Modified Teacher Drooling Scale (mTDS) score as covariate; Test type: Superiority; p = 0.032, MMRM; Least square mean (LS-mean) difference = 0.28, 95% CI 2-sided [0.02 to 0.53], Standard Error of Mean 0.127

3. Primary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs) Overall and Per Injection Cycle
Time Frame: Baseline up to Week 64
Population: SES: subset of all participants who received study medication (NT 201 or placebo) during MP or (NT 201) during OLEX of study. "n" is number of participants evaluable for this measure at a given time period and who were included in the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Number analyzed (Participants) | 72 | 148 | 35 | 214 | 33
Participants
  Overall | 11 | 27 | 5 | 92 | 15
  First injection cycle (MP): number analyzed (Participants) | 72 | 148 | 35 | 0 | 0
  First injection cycle (MP) | 11 | 27 | 5 |  |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 214 | 33
  Second injection cycle (OLEX) |  |  |  | 44 | 7
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 205 | 33
  Third injection cycle (OLEX) |  |  |  | 35 | 5
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 193 | 33
  Fourth injection cycle (OLEX) |  |  |  | 40 | 11

4. Secondary Outcome: Change From Baseline in uSFR at Weeks 8 and 12
Description: This endpoint was analyzed in double-blind, MP, 6 to 17 years participants. uSFR was assessed by weighing of absorbent swabs with safety threads soaked with saliva over 5 minutes and then procedure was repeated after 30 minutes. Salivary flow rate was equal to weight increase of swabs/time of collection. The average of the 2 results for flow rate was calculated. The reduction of measured weight over the study relates to improvement of sialorrhea.
Time Frame: Baseline and Weeks 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: g/min
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years)
Number analyzed (Participants) | 72 | 148
g/min
  Change at Week 8 | -0.07 (0.015) | -0.16 (0.012)
  Change at Week 12 | -0.06 (0.016) | -0.16 (0.013)
Statistical Analysis 1: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); Statistical analysis at Week 8: LS-Mean is from a MMRM analysis with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline uSFR score as covariate; Test type: Superiority; p < 0.0001, MMRM; Least square mean (LS-mean) difference = -0.09, 95% CI 2-sided [-0.12 to -0.05], Standard Error of Mean 0.019
Statistical Analysis 2: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); Statistical analysis at Week 12: LS-Mean is from a MMRM analysis with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline uSFR score as covariate; Test type: Superiority; p < 0.0001, MMRM; Least square mean (LS-mean) difference = -0.1, 95% CI 2-sided [-0.14 to -0.06], Standard Error of Mean 0.021

5. Secondary Outcome: GICS at Weeks 8 and 12
Description: This endpoint was analyzed in double-blind, MP, 6 to 17 years participants. The GICS was used to measure the carer's/parent's impression of change due to treatment. The response option was a common 7-point Likert scale with the following values: +3 (very much improved); +2 (much improved); +1 (minimally improved); 0 (no change); -1 (minimally worse); -2 (much worse); -3 (very much worse).
Time Frame: Weeks 8 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years)
Number analyzed (Participants) | 72 | 148
units on a scale
  Week 8 | 0.54 (0.096) | 0.94 (0.068)
  Week 12 | 0.47 (0.111) | 0.87 (0.073)
Statistical Analysis 1: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); Statistical analysis at Week 8: LS-Mean is from a MMRM analysis model with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline mTDS score as covariate; Test type: Superiority; p = 0.0008, MMRM; Least square mean (LS-mean) difference = 0.4, 95% CI 2-sided [0.17 to 0.63], Standard Error of Mean 0.116
Statistical Analysis 2: Comparison: Double-blind MP: Placebo (Age 6 to 17 Years) vs Double-blind, MP: NT 201 (Age 6 to 17 Years); Statistical analysis at Week 12: LS-Mean is from a MMRM analysis model with treatment group, pooled investigation sites, and age groups as fixed factors, visit*treatment as interaction term, visit as repeated factor, and baseline mTDS score as covariate; Test type: Superiority; p = 0.0026, MMRM; Least square mean (LS-mean) difference = 0.4, 95% CI 2-sided [0.14 to 0.66], Standard Error of Mean 0.132

6. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events of Special Interest (AESI) Overall and by Injection Cycle
Time Frame: Baseline up to Week 64
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Number analyzed (Participants) | 72 | 148 | 35 | 214 | 33
Participants
  Overall | 0 | 1 | 0 | 4 | 0
  First injection cycle (MP): number analyzed (Participants) | 72 | 148 | 35 | 0 | 0
  First injection cycle (MP) | 0 | 1 | 0 |  |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 214 | 33
  Second injection cycle (OLEX) |  |  |  | 3 | 0
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 205 | 33
  Third injection cycle (OLEX) |  |  |  | 1 | 0
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 193 | 33
  Fourth injection cycle (OLEX) |  |  |  | 0 | 0

7. Secondary Outcome: Occurrence of Treatment Emergent Serious Adverse Events (TESAEs) Overall and by Injection Cycle
Time Frame: Baseline up to Week 64
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Number analyzed (Participants) | 72 | 148 | 35 | 214 | 33
Participants
  Overall | 1 | 0 | 1 | 8 | 0
  First injection cycle (MP): number analyzed (Participants) | 72 | 148 | 35 | 0 | 0
  First injection cycle (MP) | 1 | 0 | 1 |  |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 214 | 33
  Second injection cycle (OLEX) |  |  |  | 3 | 0
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 205 | 33
  Third injection cycle (OLEX) |  |  |  | 5 | 0
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 193 | 33
  Fourth injection cycle (OLEX) |  |  |  | 0 | 0

8. Secondary Outcome: Occurrence of TEAEs Related to Treatment as Assessed by the Investigator Overall and by Injection Cycle
Time Frame: Baseline up to Week 64
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Number analyzed (Participants) | 72 | 148 | 35 | 214 | 33
Participants
  Overall | 0 | 2 | 1 | 10 | 0
  First injection cycle (MP): number analyzed (Participants) | 72 | 148 | 35 | 0 | 0
  First injection cycle (MP) | 0 | 2 | 1 |  |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 214 | 33
  Second injection cycle (OLEX) |  |  |  | 5 | 0
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 205 | 33
  Third injection cycle (OLEX) |  |  |  | 5 | 0
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 193 | 33
  Fourth injection cycle (OLEX) |  |  |  | 1 | 0

9. Secondary Outcome: Occurrence of TEAEs Leading to Discontinuation Overall and by Injection Cycle
Time Frame: Baseline up to Week 64
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
Number analyzed (Participants) | 72 | 148 | 35 | 214 | 33
Participants
  Overall | 1 | 1 | 1 | 4 | 0
  First injection cycle (MP): number analyzed (Participants) | 72 | 148 | 35 | 0 | 0
  First injection cycle (MP) | 1 | 1 | 1 |  |
  Second injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 214 | 33
  Second injection cycle (OLEX) |  |  |  | 2 | 0
  Third injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 205 | 33
  Third injection cycle (OLEX) |  |  |  | 2 | 0
  Fourth injection cycle (OLEX): number analyzed (Participants) | 0 | 0 | 0 | 193 | 33
  Fourth injection cycle (OLEX) |  |  |  | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 64
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Double-blind MP: Placebo (Age 6 to 17 Years) | Double-blind, MP: NT 201 (Age 6 to 17 Years) | Open-label, MP: NT 201 (Age 2 to 5 Years) | OLEX: NT 201 (Age 6 to 17 Years) | OLEX: NT 201 (Age 2 to 5 Years)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/148 | 0/35 | 0/214 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/148 | 1/35 | 8/214 | 0/33
Other Adverse Events (participants affected / at risk) | 3/72 | 3/148 | 2/35 | 34/214 | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MP: Placebo (Age 6 to 17 Years) (N=72) | Double-blind, MP: NT 201 (Age 6 to 17 Years) (N=148) | Open-label, MP: NT 201 (Age 2 to 5 Years) (N=35) | OLEX: NT 201 (Age 6 to 17 Years) (N=214) | OLEX: NT 201 (Age 2 to 5 Years) (N=33)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MP: Placebo (Age 6 to 17 Years) (N=72) | Double-blind, MP: NT 201 (Age 6 to 17 Years) (N=148) | Open-label, MP: NT 201 (Age 2 to 5 Years) (N=35) | OLEX: NT 201 (Age 6 to 17 Years) (N=214) | OLEX: NT 201 (Age 2 to 5 Years) (N=33)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (3) | 13 (16) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (4)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 2 (3)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (5)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT02270736/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02270736/SAP_000.pdf